CLINICAL TRIAL: NCT06605807
Title: Optimizing Prescribing Decisions for Hospitalized Older Adults With Chronic Conditions: Aim 3
Brief Title: Optimizing Prescribing Decisions for Hospitalized Older Adults With Chronic Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Timothy Anderson, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24070027; K76AG074878 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Prescribing Decisions; Diabetes; Multimorbidity; Hypertension; Geriatrics
Keywords: prescribing; hypertension; diabetes; geriatrics; polypharmacy; multimorbidity; hospital medicine
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinician Participants (Experimental): All clinician participants will undergo the same intervention, an educational session providing a clinical decision framework for managing older adults' chronic conditions during hospitalization.
  Interventions: Other: Clinical Decision Framework for Managing older adults' chronic conditions during hospitalization.

INTERVENTIONS:
Other: Clinical Decision Framework for Managing older adults' chronic conditions during hospitalization. — All clinicians will attend an educational session where they will be provided a clinical decision framework for management of chronic conditions in hospitalized older adults, reviewing guiding principles for managing chronic disease in the hospital, and working through case-based hypothetical examples.

SUMMARY:
The goal of this pilot clinical trial is to learn if providing a clinical decision framework for managing older adults chronic conditions during hospitalization to inpatient clinicians improves clinicians' ability to individualize chronic condition prescribing decisions for hospitalized older adults (65 and older). The main questions it aims to answer are:

* Will the clinical decision framework lead to clinicians having greater confidence to individualize discharge prescribing?
* Will clinicians using the framework discharge make fewer changes to hospitalized older adults with home diabetes and hypertension medications than they did prior to receiving the framework?
* Will older adult patients of participating clinicians will report fewer gaps in understanding of medication changes after the clinician is exposed to the framework?

Researchers will compare participating clinician survey responses and prescribing records from before and after an educational session presenting the clinical decision framework.

Participants will be asked to

* Attend a one-time educational session on the clinical decision framework
* Complete 2 electronic surveys, one before and one following the educational session.
* Agree for researchers to contact their patients, in order for patients to complete a one-time phone survey about changes made to home medications during hospitalization and quality of communication from the hospital team.

ELIGIBILITY:
Clinician Participants:

Inclusion Criteria:

1. Attending clinicians who practice on the general medicine or hospital medicine service at UPMC Presbyterian, UPMC Montefiore, UPMC Shadyside, UPMC Mercy, or UPMC Magee-Women's Hospital campuses.
2. Practicing on the general medicine or hospital medicine service. This population may include physicians with training in general internal medicine, hospital medicine, family practice, internal medicine subspecialities, as well as advance practice clinicians.

Exclusion Criteria:

1. Anticipating leaving current clinical position within next 3 months
2. Less than 4 weeks of inpatient attending service scheduled within 3 months of recruitment

Patient Participants:

Inclusion Criteria:

1. Adult aged 65 years or older who are hospitalized under the care of a participating clinician and discharged home.
2. Eligible patients must recieve at least one cardiometabolic medication change at hospital discharge (can include new medication starts, stops, or dose changes). Cardiometabolic medications include any class of antihypertensive, lipid lowering, anti-platelet, or glucose lowering medications regardless of indication for use.

Exclusion Criteria:

1. Incapacity for informed consent / unable to answer survey questions due to cognitive impairment
2. Enrolled in hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinician - Change in Prescribing Self-Efficacy | Baseline and two months post-intervention
  For each clinician participant the investigators will ask their self-efficacy to individualize blood pressure and diabetes treatment decisions for hospitalized older adults. Measured through ten 7-point Likert scale questions measured [Strongly Disagree - Strongly Agree]. Scores will be summed and range from 10 (all Strongly Disagree) to 70 (all Strongly Agree).

SECONDARY OUTCOMES:
Clinician - Change in Attitudes | Baseline and two months post-intervention
  The investigators will ask clinicians 8 questions about their attitudes towards individualizing antihypertensive and diabetes treatment decisions on a 7-point Likert scale. Individualizing antihypertensive and diabetes treatment decisions for hospitalized older adults is:
  Necessary - Unnecessary Beneficial - Harmful High-priority - Low-priority Worthless - Useful.
  Scores will be summed and range from 8 to 56.
Clinician - Discharge Prescribing | Pre-intervention and post-intervention (2 months before and 2 months after the intervention)
  For each clinician participant, the investigators will review the electronic health record for all hospitalized patients aged 65 years and older who were discharged alive under the clinician participant's care in the 2 months before and 2 months after the intervention to identify all antihypertensive and diabetes medication changes made during hospitalization. The investigators will compare the proportion of patients discharged with cardiometabolic medication changes in the 2 months prior to the intervention to the 2 months after the intervention. The investigators will examine proportion of patients receiving medication intensifications and the proportion receiving any medication change.
Patient - Change in Medication Discrepencies | Single time survey within a week of discharge from clinician participants care.
  The investigators will ask each enrolled patient how they are taking each of their cardiometabolic medications and compare their current reported medication use to the hospital discharge summary. The investigators will compare the proportion of patient participants reported a medication discrepancy (taking medication differently than hospital discharge summary) in the pre-intervention period to the post-intervention period.
Clinician - Acceptability of Clinical Decision Framework | 30 days post-intervention
  The investigators will ask clinicians if they used the clinical decision framework and 7 questions on a 7 point Likert scale (strongly disagree to strongly agree) regarding the framework's clarity, length, and whether it was useful. The investigators will ask what they liked about the framework and what would they change. The investigators will ask about facilitators and barriers to using the framework and whether they plan to keep using it. Scores will be summed and range from 7 to 49.
Clinician - Change in Intentions | Baseline and two months post-intervention
  The investigators will ask each enrolled clinician two questions to assess choice predisposition (leaning) towards individualizing blood pressure and diabetes medications prescribing decisions during hospitalization using two 7-point Likert Scales (Strongly Disagree to Strongly Agree). Scores will be summed and range from 2 (all Strongly Disagree) to 14 (all Strongly Agree).
Clinician - Change in Perceived Norms | Baseline and two months post-intervention
  The investigators will ask each enrolled clinician six questions on their perceptions on norms on individualizing blood pressure and diabetes treatment decisions for hospitalized older adults. Measured through 7-point Likert scale questions measured [Strongly Disagree - Strongly Agree]. Scores will be summed and range from 6 (all Strongly Disagree) to 42 (all Strongly Agree).
Clinician - Awareness of Evidence Base | Baseline and two months post-intervention
  The investigators will ask each enrolled clinician to respond to four questions regarding their familiarity with the evidence base for the treatment of blood pressure and diabetes while a patient is hospitalized. These will be framed as four 7-point Likert Scales (Strongly Disagree to Strongly Agree). Scores will be summed and range from 4 (all Strongly Disagree) to 28 (all Strongly Agree).
Patient - Change in Overall Hospital Experience | Baseline through two months post-intervention
  The investigators will ask each enrolled patient to rate their overall hospital experience from 0 to 10. Where 0 is I had a very poor experience and 10 is I had a very good experience. Scores will be summed from 0 to 10. The investigators will compare average scores of patients in the pre-intervention period to the post-intervention period
Patient - Change in Experience in the Hospital | Baseline through two months post-intervention
  The investigators will ask each enrolled patient a 4 question survey on communication during their hospital stay. Possible answers include never (1), sometimes (2), usually (3), and always (4). Scores will be summed from 4 to 16. The investigators will compare mean scores of patients in the pre-intervention period to the post-intervention period.
Patient - Change in Experience Leaving the Hospital | Baseline through two months post-intervention
  The investigators will ask each enrolled patient a 3 question survey on communication when they left the hospital. Possible answers include not at all (1), partly (2), quite a bit (3), completely (4), and not applicable (0). Scores will be summed from 0 to 12. The investigators will compare mean scores of patients in the pre-intervention period to the post-intervention period.
Patient - Change in Understanding of Medication Changes | Baseline through two months post-intervention
  The investigators will ask each enrolled patient their understanding of the reason for each cardiometabolic medication change made at hospital discharge and compare their understanding to the hospital discharge summary rationale to identify concordant versus discordant understanding. The investigators will compare the proportion of patients with discordant understanding of cardiometabolic medication changes in the pre-intervention period to the post-intervention period.
Patient - Change in Comprehension of Disease Monitoring | Baseline through two months post-intervention
  The investigators will ask each patient participant enrolled if the hospital discussed their blood pressure and/or provided guidance on disease monitoring (e.g. blood pressure or blood glucose) after discharge. The investigators will compare the proportion of patients reporting guidance on disease monitoring from the pre-intervention to post-intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Anderson, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No